CLINICAL TRIAL: NCT04336319
Title: An Exploratory Pilot Study Assessing the Efficacy of Fecal Microbial Transplantation for Clinical and Endoscopic Characteristics of Ileal Pouch Anal Anastomosis Patients
Brief Title: Fecal Microbial Transplantation for Ileal Pouch Anal Anastomosis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, R&D Department, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0210-18-TLV
Record Dates: First submitted 2019-06-04; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Ileal Pouch Anal Anastomosis
Keywords: POUCH; FMT; IPAA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a confirmed diagnosis of UC who underwent IPAA (Experimental): Patients who meet inclusion criteria will be enrolled and will sign an informed consent form. The study includes six visits to the IBD clinic and phone calls between visits.
  Interventions: Biological: Fecal Microbial Transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — 1. At baseline, the fecal fluid from 3 different donors, 150 ml, will be delivered via pouchoscopy after which the patient will roll in to the right lateral position and stay in that position for at least 15 minutes. Prior to the procedure, the patient will fast for 12 hours and preform two fleet enemas as preperation.
  2. FMT at 7 days and 4 weeks will be delivered via ingestion of 15 capsules containing 650 µL of fecal fluid from 3 different donors (the same three donors as at baseline).

SUMMARY:
The investigator is hypothesize that an intensive FMT regimen will have superior efficacy the treatment of inflammatory disorders of the pouch (pouchitis and CLDP).

DETAILED DESCRIPTION:
Study Design:

An open label non-controlled clinical trial.

Study population:

Patients aged 18 to 80 years with a confirmed diagnosis of UC , who underwent IPAA.

Recruitment of the study population:

Patients will be enrolled at the Pouch Clinic of the Tel Aviv Medical Center Inflammatory Bowel Disease Center and at the Department of Colorectal Surgery.

Study procedure:

The study includes six visits to the IBD clinic and phone calls between visits. At baseline, after 8 weeks and after one year of intervention, all patients will undergo pouchoscopy which will be recorded and scored for pouch endoscopic score (Appendix 2). In all three procedures, samples will be collected for future analysis.

According to their endoscopic evaluation at baseline, patients will be categorized as those with an inflamed pouch (cuff, afferent loop, pouch inlet, J-pouch, pouch outlet or pouch mid-line scare) or non inflamed pouch (irritable pouch patients) according to a pouch endoscopic score (PES) and the modified pouch disease activity index endoscopic domain (mPDAI).

Baseline pouchoscopy will include FMT, followed by capsule FMT after 1 week (15 capsules), and after 4 weeks of the study.

All patients will undergo clinical followup at week 4 of the study (mPDAI clinical domain, PCS and PGA) and a second pouchoscopy after 8 weeks.

Clinical follow up will be performed at week 12 of the study, and an annual endoscopic follow up will be preformed at 52 weeks or per personal indication.

Data collection at baseline and follow-up visits will include:

1. Clinical assessment:

   * Pouch clinical score (PCS)
   * mPDAI - clinical domains
   * Physician Global Assessment (PGA)
   * Pouch endoscopic score (PES)
2. Collection of biological samples:

   * Stool for analysis of calprotectin level and microbiome
   * Urine for analysis of metabolomics
   * Serum for analysis of complete blood count (CBC), serum levels of C-Reactive Protein (CRP), albumin, creatinine, liver enzymes
   * Tissue samples collected during pouchoscopy at baseline and followup - samples will be collected from the cuff, pouch body and pouch inlet.
3. Anthropocentric measures will be assessed (weight, height)
4. Complete study questionnaires:

   * A validated lifestyle and food frequency questionnaire (FFQ)
   * Three day food diary
   * Quality of life questionnaire (SF-12)
   * Patient-reported outcomes (PRO) Measurement Information System (PROMIS)
   * Life style questionnaire

Safety assessments:

will include history taking, vital signs, physical examinations and laboratory analysis during each visit. Patients who discontinue the trial treatment will continue to be followed as per protocol. Follow-up will be discontinued in patients who withdraw informed consent or are lost for follow-up. All adverse events will be registered as: unrelated, possible related, likely related or definitely related to the intervention. SAEs will be communicated immediately to the IRB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years with a confirmed diagnosis of UC, who underwent IPAA.
2. Endoscopic deterioration or Clinically suspected pouchitis, defined as increased bowel frequency (≥1 stools) relative to post-IPAA baseline (1-3 months post IPAA).
3. Clinically stable patients on constant medical regimen throughout the study period. Treated by mesalamine for at least 6 weeks, or steroids at least 2 week, or immunomodulator or biologic at least 12 weeks, medical cannabis at least 2 weeks

Exclusion Criteria:

1. Diagnosis of Crohn's disease or indeterminate colitis prior to IPAA.
2. Positive stool test for parasites or stool culture for pathological bacteria within 60 days prior to enrollment.
3. Evidence or history of Clostridium difficile infection within 60 days prior to enrollment.
4. Active clinically significant infection (within 60 days of enrollment).
5. Active septic pouch complication (e.g., abscess, leak, fistula).
6. Post-surgical complication of the pouch (e.g., obstruction, stricture, volvulus, prolapse).
7. Pregnancy or lactation.
8. Unstable or uncontrolled medical disorder (other than suspected pouchitis).
9. Inability to give informed consent and complete the study protocol.
10. Patient participating in other concomitant clinical intervention trial or who had received any experimental drug within a month prior to enrollment
11. Patients received antibiotics within 2 days of enrollment, or are anticipated to use antibiotics or probiotics within the study period (elective surgery or dental care).
12. Patients received fecal transplantation in the last 6 months.
13. Fever>38°c
14. An active malignant disease or a prior malignancy during the previous 5 years (excluding skin BCC).
15. Inability or reluctance to follow through with the study protocol, including (but not exclusive) to: colonoscopy, enema, study visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
safety of fecal microbial transplantation in pouch patients by disease exacerbations | 1 year
  determine whether manipulation of gut microbiome by FMT to IPAA patients is safe safety of FMT will be measured by rate of patients with disease exacerbations
safety of fecal microbial transplantation in pouch patients by hospitalizations of patients | 1 year
  determine whether manipulation of gut microbiome by FMT to IPAA patients is safe safety of FMT will be measured by amount of patients that require hospitalizations
safety of fecal microbial transplantation in pouch patients by patients requiring surgery | 1 year
  determine whether manipulation of gut microbiome by FMT to IPAA patients is safe safety of FMT will be measured by amount of patients that require surgery
efficacy of FMT in pouch patients measured by mPDAI decrease | 2 months
  By preforming a pouchoscopy, mPDAI (modified pouchitis disease activity index) will be used to assess decrease of ≤1 in mPDAI in condition of the pouch comparing to baseline
efficacy of FMT in pouch patients measured by clinical remission | 2 months
  efficacy of FMT in pouch patients will be measured by the amount of patients with clinical remission measured by mPDAI clinical score <3

SECONDARY OUTCOMES:
efficacy of FMT in pouch patients measured by amount of patients with sustained remission | 12 months
  Sustained remission as defined by mPDAI endoscopic score ≤ 1 or mPDAI endoscopic and clinical ≤ 5
efficacy of FMT in pouch patients measured by amount of patients with sustained clinical remission | 12 months
  Sustained remission as defined by mPDAI clinical <3
efficacy of FMT in pouch patients measured by reduce of inflammatory markers | 1 month
  Reduction in inflammatory markers (calprotectin and CRP)
efficacy of FMT in pouch patients measured by reduce of inflammatory markers | 2 months
  Reduction in inflammatory markers (calprotectin and CRP)
efficacy of FMT in pouch patients measured by reduce of inflammatory markers | 3 months
  Reduction in inflammatory markers (calprotectin and CRP)
efficacy of FMT in pouch patients measured by reduce of inflammatory markers | 12 months
  Reduction in inflammatory markers (calprotectin and CRP)
efficacy of FMT in pouch patients measured by reduce of PGA (physical global assessment) | 1 month
  Reduction in PGA (physical global assessment) comparing to baseline
efficacy of FMT in pouch patients measured by reduce of PGA (physical global assessment) | 2 months
  Reduction in PGA (physical global assessment) comparing to previous assessments
efficacy of FMT in pouch patients measured by reduce of PGA (physical global assessment) | 3 months
  Reduction in PGA (physical global assessment) comparing to previous assessments
efficacy of FMT in pouch patients measured by reduce of PGA (physical global assessment) | 12 months
  Reduction in PGA (physical global assessment) comparing to previous assessments
efficacy of FMT in pouch patients measured by improvement of life quality | 1 month
  efficacy of FMT by filling questionnaire describing life quality and comparing to baseline to observe improvement
efficacy of FMT in pouch patients measured by improvement of life quality | 2 months
  efficacy of FMT by filling questionnaire describing life quality and comparing to baseline to observe improvement
efficacy of FMT in pouch patients measured by improvement of life quality | 3 months
  efficacy of FMT by filling questionnaire describing life quality and comparing to baseline to observe improvement
efficacy of FMT in pouch patients measured by improvement of life quality | 12 months
  efficacy of FMT by filling questionnaire describing life quality and comparing to baseline to observe improvement
efficacy of FMT in pouch patients measured by improvement of nutritional status | 1 month
  improvement of patients nutritional status comparing to baseline measured by BMI (body Mass Index). Normal range is BMI of 18.5-25
efficacy of FMT in pouch patients measured by improvement of nutritional status | 2 months
  improvement of patients nutritional status comparing to baseline measured by BMI (body Mass Index). Normal range is BMI of 18.5-25
efficacy of FMT in pouch patients measured by improvement of nutritional status | 3 months
  improvement of patients nutritional status comparing to baseline measured by BMI (body Mass Index). Normal range is BMI of 18.5-25
efficacy of FMT in pouch patients measured by improvement of nutritional status | 12 months
  improvement of patients nutritional status comparing to baseline measured by BMI (body Mass Index). Normal range is BMI of 18.5-25

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No